CLINICAL TRIAL: NCT02980848
Title: Comparative Effectiveness of Breast Cancer Screening and Diagnostic Evaluation by Extent of Breast Density
Brief Title: Assessing Breast Density's Value in Imaging - A Comparative Effectiveness Study
Acronym: BCSC-ADVANCE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of California, Davis (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of California, San Francisco (Other); Dartmouth College (Other); Kaiser Permanente (Other); University of Vermont (Other); University of North Carolina (Other); University of Illinois at Chicago (Other); Wake Forest University Health Sciences (Other); Harvard Pilgrim Health Care (Other); Albert Einstein College of Medicine (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 941466; PCS-1504-30370 (Other: PCORI)
Record Dates: First submitted 2016-11-19; First posted 2016-12-02 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: digital mammography; digital breast tomosynthesis; breast magnetic resonance imaging; screening; breast density; breast imaging; pre-operative magnetic resonance imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screening group: Women without a history of breast cancer undergoing screening digital mammography, screening digital breast tomosynthesis, or screening breast magnetic resonance imaging.
  Interventions: Other: Screening digital mammography; Other: Screening digital breast tomosynthesis; Other: Screening breast magnetic resonance imaging
- Women with breast cancer: Women diagnosed with stage 0-III breast cancer undergoing pre-operative work-up with diagnostic mammography alone or diagnostic mammography plus pre-operative breast magnetic resonance imaging.
  Interventions: Other: Diagnostic mammography; Other: Pre-operative breast magnetic resonance imaging

INTERVENTIONS:
Other: Screening digital mammography — Screening with digital mammography alone
  Groups: Screening group
Other: Screening digital breast tomosynthesis — Screening with digital mammography plus digital breast tomosynthesis
  Groups: Screening group
Other: Screening breast magnetic resonance imaging — Screening with digital mammography plus breast magnetic resonance imaging
  Groups: Screening group
Other: Diagnostic mammography — Pre-operative diagnostic work-up with mammography alone
  Groups: Women with breast cancer
Other: Pre-operative breast magnetic resonance imaging — Pre-operative diagnostic work-up with mammography plus breast magnetic resonance imaging
  Groups: Women with breast cancer

SUMMARY:
This Breast Cancer Surveillance Consortium (BCSC) ADVANCE study is a large, observational pragmatic comparative effectiveness research study using high-quality, prospectively collected data from BCSC registries to generate evidence on how breast density should be integrated into decision making around breast cancer screening and preoperative diagnostic work-up. We will augment existing BCSC registry infrastructure with additional prospective data collection and collection of patient reported outcomes (PROs), CISNET modeling of long-term screening outcomes, and qualitative data from focus groups with women represented in two aims.

DETAILED DESCRIPTION:
Aim 1: Compare the effectiveness of breast cancer screening using digital mammography alone versus digital mammography plus supplemental screening (digital breast tomosynthesis or MRI) by extent of breast density.

Sub aim 1: Evaluate whether the performance of tomosynthesis improves with years of experience, and whether any "learning curve" depends on radiologist specialty (i.e., breast imaging specialist vs. general radiologist).

Aim 2: Compare the effectiveness of preoperative MRI versus no MRI by extent of breast density among women with an initial, pathologically confirmed diagnosis of DCIS or invasive breast cancer.

Covid-19 Enhancement Aim and Hypotheses:

Develop patient-focused messaging content through focus groups that radiology facilities can use when scheduling appointments to inform women of the safety to schedule or postpone breast screening or diagnostic services.

ELIGIBILITY:
Aim 1 Clinical Outcomes

Inclusion criteria:

* Women aged 40-79 undergoing screening mammography from 2010-2017 for comparisons with tomosynthesis and 2005-2017 for comparison with breast MRI at a facility that participates in one of six BCSC breast imaging registries
* Digital mammography exams performed for screening and performed with or without supplemental screening with digital breast tomosynthesis from 2010-2017 or breast MRI from 2005-2017, at a facility that participates in one of seven BCSC breast imaging registries, and in women who meet inclusion criteria.

Exclusion criteria:

* Exams performed on women with a history of breast cancer, mastectomy, or breast augmentation.
* Unilateral mammograms and mammograms performed within 9 months of a prior mammogram to avoid classifying diagnostic exams as screening
* Exams without complete cancer capture during the follow-up period

Aim 1 Patient Reported Outcomes

Inclusion criteria:

* Women aged 40-74 years undergoing screening mammography, with or without supplemental screening with digital breast tomosynthesis or breast MRI, at selected BCSC facilities
* Women within 12 months of a digital screening mammogram with known breast density and no known breast cancer diagnosis
* For MRI subgroup, we will include women with a screening MRI within the prior 24 months
* Within strata defined by BCSC registry, breast density subgroup (dense vs. not dense), and race/ethnicity, women with supplemental screening with digital breast tomosynthesis or breast MRI will be matched to women without supplemental screening

Aim 1 Focus Groups

Inclusion criteria:

* Women age 40-74 years undergoing screening mammography, with or without supplemental screening (defined as digital breast tomosynthesis or breast MRI)
* Women within 12 months post-most recent screening examination with known dense breasts from most recent screening mammogram and no known breast cancer diagnosis
* Women who are able to speak English and can travel to a nearby location for a discussion

Subaim 1

Inclusion criteria:

* Radiologists interpreting digital mammography and/or tomosynthesis for at least one year from 2010-2017 at a facility that participates in the BCSC
* Digital mammography exams and digital breast tomosynthesis performed for screening and evaluated by a radiologist meeting inclusion criteria from 2010-2017

Exclusion criteria:

* Exams performed on women with a history of breast cancer, mastectomy, or breast augmentation
* Unilateral mammograms and mammograms performed within 9 months of a prior mammogram to avoid classifying diagnostic exams as screening
* Exams without complete cancer capture during one year following the screening mammogram

Aim 2 Clinical Outcomes

Inclusion criteria:

* Women at least 18 years of age with a first breast cancer diagnosis (DCIS or invasive) from 2005-2017 for whom there was a mammogram performed within the year prior to breast cancer diagnosis at one of the participating BCSC registry facilities
* Women for whom we have pathologically-confirmed breast cancer (DCIS or invasive) with a pathology or biopsy record related to the incident cancer diagnosis in the BCSC data
* MRI and mammography examinations performed for pre-operative work-up from 2005-2017 at one of the participating BCSC registry facilities in women meeting eligibility criteria

Aim 2 Patient Reported Outcomes

Inclusion criteria:

* Women at least 18 years of age with a first pathology-confirmed breast cancer diagnosis (DCIS or stage I-III invasive) within 6-18 months
* Known breast density at the time of breast cancer diagnosis

Aim 2 Focus Groups

Inclusion criteria:

* Women age ≥18 with a first breast cancer diagnosis (DCIS or stage I-III invasive cancer) within 1-5 years and after completion of active breast cancer treatment who have undergone mammography or MRI pre-operatively.
* Women who are able to speak English and can travel to a nearby location for a discussion

COVID-19 Enhancement Focus Groups

Inclusion criteria:

* Women age 18-74 who were due for breast imaging services during the COVID pandemic and have either canceled their appointment, delayed their appointment, or kept their appointment
* Women who are able to speak English and can attend calls virtually through Zoom or over the phone
* In addition, for focus groups with women who have prior breast cancer:

  1. First breast cancer diagnosis (DCIS or stage I-III invasive cancer) within 1-3 years prior to March, 2020.
  2. Completed active cancer treatment (ongoing endocrine and Herceptin therapy acceptable)
  3. No evidence of a second breast cancer event in cancer registry or pathology data before recruitment.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include women age 40-79 undergoing screening mammography (Aim 1) and women age ≥18 with a first breast cancer diagnosis (Aim 2). We will include women in the BCSC cohort with mammography from 2005-2017. BCSC participants are identified from seven BCSC breast imaging registries. The BCSC prospectively collects data during routine clinical practice through voluntary partnerships with radiology facilities. Women enter the BCSC cohort when they receive a breast-imaging exam at a participating facility.
Sampling Method: Non-Probability Sample
Enrollment: 1341172 (Actual)
Dates: Start 2016-09; Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Screening Benefits: Rate of early stage invasive cancer detection (Aim 1) | Within one year after screen
  Number of stage I or IIA cancers diagnosed within 1 year of a positive screen divided by total number of screens
Screening Failures: Interval or advanced breast cancer rate (Aim 1) | Within one year after screen
  Number of invasive cancer cases within 1 year of a negative screen divided by total number of screens
  Number of advanced cancers (stage IIB or higher) within 1 year of a screen divided by total number of screens
Screening Harms: Recall rate (Aim 1) | Within one year after screen
  Number of positive screens divided by total number of screens
Screening Harms: False-positive (FP) recall rate (Aim 1) | Within one year after screen
  Number of positive screens without a cancer diagnosed within 1 year divided by total number of screens
Screening Harms: FP biopsy recommendation rate (Aim 1) | Within one year after screen
  Number of screens with a biopsy recommendation and no cancer diagnosed within 1 year divided by total number of screens
Screening Harms: Other consequences (Aim 1) | Within one year after screen
  Number of DCIS diagnoses within 1 year of a positive screen divided by total number of screens, reported overall and by grade
Patient Reported Outcomes (Aim 1) | Measured within one year post-screening
  Patient surveys targeted to determining outcomes of interest to patients
Rates of additional breast cancers detected (Aim 2) | 6 months after initial diagnosis
  Number of women with contralateral breast cancer diagnosed within 6 months of initial diagnosis over total number of women
3-year rate of 2nd breast cancer events (Aim 2) | 3 years after initial diagnosis
  Rate of 2nd breast cancers diagnosed within 3 years of follow-up (starting 6 months after initial diagnosis) calculated separately for ipsilateral and contralateral cancers
Patient Reported Outcomes (Aim 2) | Measured 6-18 months post-diagnosis
  Patient surveys targeted to determining outcomes of interest to patients

SECONDARY OUTCOMES:
Performance Measures: Sensitivity (Aim 1) | Within one year after screen
  Number of cancer cases within 1 year of positive screen divided by number of breast cancer cases
Performance Measures: Specificity (Aim 1) | Within one year after screen
  Number of negative screens without cancer diagnosed within 1 year of screen divided by number of screens without breast cancer
Performance Measures: Positive predictive value (Aim 1) | Within one year after screen
  Number of cancer cases within 1 year of positive screen divided by number of positive screens
Definitive surgery type (Aim 2) | 6 months after initial diagnosis
  Rates of unilateral mastectomy, or bilateral mastectomy, lumpectomy with reconstruction, lumpectomy without reconstruction
Negative predictive value of work-up with MRI (Aim 2) | 6 months after initial diagnosis
  Number of women with a negative pre-operative MRI and no additional cancers diagnosed within 6 months after initial diagnosis over the total number of women with a negative pre-operative MRI
Negative predictive value of work-up without MRI (Aim 2) | 6 months after initial diagnosis
  Number of women without a pre-operative MRI with no additional cancers diagnosed within 6 months after initial diagnosis over the total number of women without a pre-operative MRI
Core biopsy rates (Aim 2) | 6 months after initial diagnosis
  Number of core biopsies within 6 months of initial diagnosis over number of breast biopsies
Surgical biopsy rate (Aim 2) | 6 months after initial diagnosis
  Number of surgical biopsies within 6 months of initial diagnosis over number of breast biopsies
Benign biopsy rate (Aim 2) | 6 months after initial diagnosis
  Number of initial benign biopsies over number of breast biopsies

OTHER OUTCOMES:
Modeled Long-Term Mortality Outcome: Breast cancers deaths averted (Aim 1) | From date of first screening examination until the date of death from any cause, up to 100 years of age
  Breast cancers deaths averted estimated by the Cancer Intervention and Surveillance Modeling Network (CISNET) models
Modeled Long-Term Mortality Outcome: Life-years gained (Aim 1) | From date of first screening examination until the date of death from any cause, up to 100 years of age
  Life-years gained estimated by the Cancer Intervention and Surveillance Modeling Network (CISNET) models
Modeled Long-Term Mortality Outcome: Overdiagnosis (Aim 1) | From date of first screening examination until the date of death from any cause, up to 100 years of age
  Overdiagnosis estimated by the Cancer Intervention and Surveillance Modeling Network (CISNET) models

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Miglioretti, PhD, Principal Investigator — University of California, Davis
Locations (7):
- United States (7):
  - Sacramento Area Breast Imaging Registry, Davis, California
  - San Francisco Mammography Registry, San Francisco, California
  - Metro Chicago Breast Cancer Registry, Chicago, Illinois
  - New Hampshire Mammography Network, Lebanon, New Hampshire
  - Carolina Mammography Registry, Chapel Hill, North Carolina
  - Vermont Breast Cancer Surveillance System, Burlington, Vermont
  - Kaiser Permanente Washington Breast Cancer Surveillance Registry, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Please visit http://www.bcsc-research.org for information about requesting BCSC data.

REFERENCES:
- [Derived] Smith RE, Sprague BL, Henderson LM, Kerlikowske K, Miglioretti DL, Wernli KJ, Onega T, diFlorio-Alexander RM, Tosteson ANA. Breast density knowledge and willingness to delay treatment for pre-operative breast cancer imaging among women with a personal history of breast cancer. Breast Cancer Res. 2024 Apr 29;26(1):73. doi: 10.1186/s13058-024-01820-x. PMID 38685119
- [Derived] Tosteson ANA, Schifferdecker KE, Smith RE, Wernli KJ, Zhao W, Kaplan CP, Buist DSM, Henderson LM, Sprague BL, Onega T, Budesky J, Jackson-Nefertiti G, Johnson D, Miglioretti DL, Kerlikowske K. Women's Breast Cancer Screening Confidence by Screening Modality and Breast Density: A Breast Cancer Surveillance Consortium Survey Study. J Womens Health (Larchmt). 2022 Nov;31(11):1547-1556. doi: 10.1089/jwh.2021.0649. PMID 36356184
- [Derived] Onega T, Zhu W, Kerlikowske K, Miglioretti DL, Lee CI, Henderson LM, Tosteson ANA, Wernli KJ, diFlorio R, Weaver DL, Buist DSM. Preoperative MRI in breast cancer: effect of breast density on biopsy rate and yield. Breast Cancer Res Treat. 2022 Jan;191(1):177-190. doi: 10.1007/s10549-021-06418-x. Epub 2021 Oct 22. PMID 34686934
- See also: Breast Cancer Surveillance Consortium (BCSC) — https://www.bcsc-research.org/